CLINICAL TRIAL: NCT00635921
Title: Ziprasidone in the Treatment of Borderline Personality Disorder: A Double-Blind, Placebo-Controlled, Randomized Study
Brief Title: Ziprasidone in the Treatment of Borderline Personality Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Ministry of Health, Spain (Other Government); REM-TAP Network (Unknown); Pfizer (Industry)
Responsible Party: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Víctor Pérez Sola
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSP-2003-002; HSP-2003-002
Record Dates: First submitted 2008-03-11; First posted 2008-03-14 (Estimated); Last update posted 2008-03-14 (Estimated); Status verified 2008-03

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder; ziprasidone
MeSH Terms: conditions — Borderline Personality Disorder | interventions — ziprasidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I ziprasidone (Active Comparator)
  Interventions: Drug: ziprasidone
- II placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ziprasidone — Dose flexible from 40 to 200 mg/d during 12 weeks
  Arms: I ziprasidone
Drug: Placebo — flexible doses from 40 to 200 mg/d during 12 weeks
  Arms: II placebo

SUMMARY:
Objective: The aim of this double-blind, placebo-controlled study was to evaluate the efficacy and tolerability of ziprasidone in the treatment of adult patients with Borderline Personality Disorder (BPD).

Method: Sixty BPD patients were included in a 12-week, single-center, double-blind, placebo-controlled study. The subjects were randomly assigned to ziprasidone or placebo in a 1:1 ratio following a two-week baseline period. The Clinical Global Impression scale for use in BPD patients (CGI-BPD) was the primary outcome measure, and other scales and self-reports related to affect, behavior, psychosis, general psychopathology domains and clinical safety were included.

DETAILED DESCRIPTION:
The American Psychiatric Association (APA) Guidelines for the Treatment of Borderline personality disorder recommend that pharmacological treatment for BPD has an important adjunctive role, especially for diminution of symptoms such as affective instability, impulsivity, psychotic-like symptoms, and self-destructive behavior. Studies conducted with low doses of conventional antipsychotics have showed significant improvements in specific symptoms such as hostility, impulsiveness, mood, and psychotic symptoms.

The introduction of atypical antipsychotics, with a more favorable tolerance profile, increases clinicians' options for treating BPD. Olanzapine has proven its efficacy in four double-blind, placebo-controlled clinical trials in patients with BPD. Ziprasidone is an atypical antipsychotic with a pharmacological action on serotonergic, dopaminergic and adrenergic receptors. It has proven to be effective for schizophrenia, schizoaffective and acute mania disorders and the incidence of side effects is low.

Although clinical findings and the pharmacological activity of ziprasidone suggest the drug may have therapeutic benefits in BPD patients, no controlled studies have yet been conducted in these patients. We carried out a randomized, double-blind, placebo-controlled study to evaluate efficacy and tolerability of ziprasidone in the management of BPD patients with moderate-high clinical severity.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of Borderline Personality Disorder
* Age between 18 and 45 years
* Clinical Global Impression of Severity (CGI-S)scores >4

Exclusion Criteria:

* No comorbidity with schizophrenia, drug-induced psychosis, organic brain syndrome, alcohol or other substance dependence, bipolar disorder, mental retardation, or major depressive episode in course
* current use of medically accepted contraception in the case of female patients.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2004-03; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
CGI scale for use in borderline personality disorder (CGI-BPD) | 12 weeks

SECONDARY OUTCOMES:
Hamilton Rating Scale Depression (HAM-D-17) | 12 weeks
Hamilton Rating Scale for Anxiety (HAM-A) | 12 weeks
Brief Psychiatric Rating Scale (BPRS) | 12 weeks
SCL-90-R | 12 weeks
Barratt Impulsiveness Scale | 12 weeks
Treatment-emergent adverse events | 12 weeks
UKU Side Effect Rating Scale | 12 weeks
EKG and laboratory assessment | 12 weeks
Buss-Durkee Inventory | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, Sta. Creu and St. Pau Hospital, Barcelona, Spain

REFERENCES:
- [Derived] Stoffers-Winterling JM, Storebo OJ, Pereira Ribeiro J, Kongerslev MT, Vollm BA, Mattivi JT, Faltinsen E, Todorovac A, Jorgensen MS, Callesen HE, Sales CP, Schaug JP, Simonsen E, Lieb K. Pharmacological interventions for people with borderline personality disorder. Cochrane Database Syst Rev. 2022 Nov 14;11(11):CD012956. doi: 10.1002/14651858.CD012956.pub2. PMID 36375174
- [Derived] Pascual JC, Soler J, Puigdemont D, Perez-Egea R, Tiana T, Alvarez E, Perez V. Ziprasidone in the treatment of borderline personality disorder: a double-blind, placebo-controlled, randomized study. J Clin Psychiatry. 2008 Apr;69(4):603-8. doi: 10.4088/jcp.v69n0412. PMID 18251623